CLINICAL TRIAL: NCT02585193
Title: Evaluation of a Commercial Program on Weight Loss and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Renee J. Rogers, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO15040047
Record Dates: First submitted 2015-10-12; First posted 2015-10-23 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight Watchers Intervention (Other): All participants are enrolled in this single arm of the study. All participants receive the Weight Watchers intervention which consists of weekly group intervention/support meetings in which weight loss behaviors (diet, physical activity) are discussed.
  Interventions: Behavioral: Weight Watchers Intervention

INTERVENTIONS:
Behavioral: Weight Watchers Intervention — All participants are enrolled in this single arm of the study. All participants receive the Weight Watchers intervention which consists of weekly group intervention/support meetings in which weight loss behaviors (diet, physical activity) are discussed.

SUMMARY:
While some evidence on weight change elicited from commercially available weight loss programs, such as Weight Watchers, is available, there is little evidence evaluating any health-related outcomes that result from losing weight through these programs. In addition, little data exists on the adherence and satisfaction of these types of programs. The purpose of this study is to evaluate body weight and health-related outcomes that are achieved from participating in a Weight Watchers program, along with program adherence and satisfaction. Men and women (N=150) that are participating in Weight Watchers weight loss program will undergo assessments at the University of Pittsburgh to evaluate outcomes related to the Weight Watchers 6 month intervention. Assessment visits, separate from the intervention, will take place at baseline (0 months), 3 months and 6 months for approximately 90 minutes at the Physical Activity and Weight Management Research Center. Participants will be asked to undergo assessments of body weight, height, aerobic stamina, functional fitness, flexibility, and complete a series of questionnaires related to demographics, program satisfaction, sleep quality, happiness, and food cravings. Adherence to the program will be measured by the number of group sessions attended.

DETAILED DESCRIPTION:
There is a body of evidence that has evaluated the effect of Weight Watchers, a commercially available weight loss program, on changes in body weight. The current investigation aims to add to this body of evidence by providing additional data on changes in body weight and enhance the current evidence-base in regards to evaluating other health-related outcomes.

There is no evidence that demonstrates whether or not the weight loss as a result of the Weight Watchers program elicits changes in health-related outcomes related to aerobic capacity, flexibility, functional fitness, sleep, and other psychological measures. Additionally, within a scientific research protocol, measures of adherence and satisfaction have not been evaluated. This study will evaluate these outcomes beyond weight changes achieved across the 24-week program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over age 18. Set "soft quotas" on the number of male and female participants - The desire is to have a 90% female / 10% male split.
* With or without previous Weight Watchers experience. Set quota on the number of participants with previous Weight Watchers experience at 65%.
* Self reported height/weight resulting in a Body Mass Index (BMI) of 27 to 43 kg/m2 (will re-screen at facility).
* Self report that he/she feels the need to lose weight.
* Willing to discontinue any current over-the-counter (OTC) supplements not recommended/prescribed by physician, with the exception of multivitamins or other vitamin supplement.
* Willing to follow recommendations required by study protocol.
* Willing to include demographic information (e.g., ethnicity, income and education).
* Willing to participate in consumer surveys and focus groups as a part of the intervention.
* Use of a personal smartphone on a daily basis. For Android devices, must be version 4.4 (code: KitKat) or 5.0 (codename: Lollipop). For iPhones, must be iOS6 and above. Cannot accommodate Blackberry devices.
* The willingness and ability to navigate and use applications on their smartphone on a daily basis (minimum training will be provided).
* Reliable home WiFi access
* Ability to commit to attending up to 27 study visits in approximately 26 weeks:

  * Ability to commit (to best of their ability) to attending weekly meetings, 30-60 minutes in duration, at the same day and time each week for 24 consecutive weeks (daytime and evening options will be available).
  * Ability to commit to up to 3 additional study visits at Weeks 0, 12, and 24, each approximately 90 minutes in duration, to complete assessments (height, weight, questionnaires, physical measures).

Exclusion Criteria:

* Participants that are currently following a commercial weight-loss program.
* Participants that have been involved in a related market research program within the last 6 months.
* Pregnant or nursing, or planning on becoming pregnant over the next 9 months.
* Recent weight loss of ≥ 5 kg in the previous 3 months.
* History of clinically diagnosed eating disorder.
* Orthopedic limitations preventing participation in regular physical activity.
* Untreated thyroid disease or > 1 change in dose or type of thyroid medication over previous 6 months.
* Taking any prescription medication with known effects on appetite or weight.

  *With the exception of subjects on a stable dose of SSRIs (Selective Serotonin Re-uptake Inhibitors) for 6 months.
* Taking oral steroids.
* Chronic/inflammatory gastrointestinal disorders (irritable bowel syndrome acceptable).
* Previous surgical procedure for weight loss.
* Major surgery within the previous 3 months.
* History of heart problems (e.g., angina, bypass surgery, MI, etc) within previous 3 months.
* Presence of implanted cardiac defibrillator or pacemaker.
* Uncontrolled hypertension self-reported BP > 160/100mmHg)
* Diuretic use for hypertension over 1.5mg per day
* Diagnosis of type 1 or type 2 diabetes
* History of presence of cancer (completely respected basal or squamous cell carcinoma acceptable if treatment completed more than 6 months prior to enrollment).
* Consuming more than 14 alcoholic drinks per week or not more than 3 drinks per day.
* Planning to relocate in the next 9 months
* Any orthopedic limitation preventing participation in regular physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Body Weight Change | 6 months
  To examine the effect of a 24-week commercially available weight loss program on weight change.

SECONDARY OUTCOMES:
Change in Sleep Quality and Duration | 6 months
  Sleep quality and duration. Participants will be asked to complete the Pittsburgh Sleep Quality Index (PSQI) at baseline, Months 3 and 6. The PSQI is a validated self-report measure of sleep duration and sleep quality.
Change in Happiness | 6 months
  Participants will be asked to complete the Oxford Happiness Questionnaire at baseline, Months 3 and 6. The OHQ is a validated self-report measure for broad personal happiness. Respondents rate 29 sentences on a 6 point Likert scale (1, strongly disagree; 6, strong agree).
Change in Food Cravings | 6 months
  The Food Craving Inventory-II (FCI-II) is a validated self-report measure for general cravings and cravings for specific types of foods and will be completed at baseline, Months 3 and 6. Respondents rate the frequency of cravings since the last time they completed the survey for each of 33 food items using a five-point Likert scale (1, never; 2, rarely; 3, sometimes; 4, often; 5, always/almost every day). The FCI-II consists of 5 scales (sweets, high fats, carbohydrates/starches, fast food fats, and fruits & vegetables) that constitute the higher order construct of food cravings (the total score).
Program Satisfaction | 6 months
  Program Satisfaction. Two parts to evaluate:
  1. Satisfaction Survey. Participants will be asked to complete a program Satisfaction Survey. The Satisfaction Survey is a self-administered survey scored on a 5-point Likert scale.
  2. Open-ended Satisfaction Survey. Participants will be asked to complete a Open-ended Satisfaction survey that consist of 2 open-ended questions, and asked respondents to report on their satisfaction with the dietary plan.
Program Adherence | 6 months
  Data on adherence (attendance at meetings and use of the points system) will also be collected. Attendance data will be recorded by Weight Watchers staff at every meeting. These data will be confirmed by a member of the research staff that will be attending the weekly Weight Watchers meetings. In addition, the weekly weights obtained at the intervention sessions will be provided to the investigators by the intervention staff to allow for examination of the trajectory of weight loss.
Change in Aerobic Capacity, Functional Fitness, Balance, Flexibility | 6 months
  Aerobic Capacity: Participants will complete a 6 minute walk test on a designated walking course. The 6 minute walk test is a measure of functional and aerobic capacity. Participants will asked to walk at a brisk, yet comfortable pace for a total of 6 minutes.
  Functional Fitness and Balance: The Short Physical Performance Battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests to measure functional fitness.
  Flexibility: Lower body flexibility will be assessed through the sit and reach test. The sit and reach is a common test to measure lower back and lower body flexibility. This will be collected 3 times with the best of 3 scores utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Renee J Rogers, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Physical Activity and Weight Management Research Center / University of Pittsburgh, Pittsburgh, Pennsylvania, United States